CLINICAL TRIAL: NCT02780102
Title: Comparison of the Effects of Cognitive-Motor Rehabilitation, Stimulant Drugs, and Active Control on Executive Functions and Clinical Symptoms of Attention Deficit/ Hyperactivity Disorder
Brief Title: Cognitive-Motor Rehabilitation, Stimulant Drugs, and Active Control in the Treatment of ADHD
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allameh Tabatabai University (Other)
Responsible Party: Principal Investigator, Saeed Azami, Mr., Allameh Tabatabai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 328/94/16090
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Cognitive-motor rehabilitation; Active Control Group; Stimulant Medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive-Motor Rehabilitation (Experimental): Cognitive-Motor Rehabilitation (CMR): 20 sixty-minute sessions of cognitive-motor rehabilitation
  Interventions: Other: Cognitive-Motor Rehabilitation
- Ritalin (Experimental): 2 to 3 doses of 10 mg Ritalin tablets per day during 8 week.
  Interventions: Drug: Ritalin
- Active Control (Active Comparator): Active Control group simultaneously received 20 sixty-minute sessions of low dose cognitive-motor exercises
  Interventions: Other: Active Control

INTERVENTIONS:
Other: Cognitive-Motor Rehabilitation — Cognitive-Motor Rehabilitation (CMR) group received 20 sixty-minute sessions of cognitive-motor exercises
  Arms: Cognitive-Motor Rehabilitation
Drug: Ritalin — 2 or 3 doses of 10 mg tablets of immediate-release Methylphenidate (Ritalin) per day for 8 week.
  Other Names: drug therapy
  Arms: Ritalin
Other: Active Control — Active Control group simultaneously received 20 sixty-minute sessions of low dose cognitive-motor exercises
  Arms: Active Control

SUMMARY:
The investigators administered a randomized controlled trial (RCT) through random assignment of children with ADHD into three different groups to compare the effects of cognitive-motor rehabilitation, immediate release methylphenidate, and an active control on the executive functioning, learning, and behavioral symptoms of children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Receiving ADHD diagnosis
* aged between 9 and 12 years
* Intelligence Quotient (IQ)>90

Exclusion Criteria:

* Severe co-morbid disorders, such as depression, op-positional defiant disorder and conduct disorder
* A history of seizures during past 2 years
* Disability or handicap preventing the child from participating cognitive-motor exercises
* Sever medical conditions requiring immediate medical treatment

Ages: 9 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Forward/backward digit span tasks from the Wechsler intelligence scale for children 4th edition (WISC-IV) | 12 months
Span board task from the Lumosity.com online brain training software | 12 months
Listening span task (L.SPAN) | 12 months
Stroop color-word test | 12 months
Tower of London test (TOL) | 12 months
Restricted academic situation scale (RASS) | 12 months
Arithmetic task from WISC-IV testing battery | 12 months
Swanson, Nolan, and Pelham's parent rating scale (SNAP-IV) | 12 months
Dictation and Spelling examination | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Azami, PhD, Study Director — Semnan University; Zeynab AliMadadi, MD, Principal Investigator — Tehran University of medical Science
Locations (1):
- Counseling and guidence Center of the Department of education of region 9 of Tehran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No